CLINICAL TRIAL: NCT05221099
Title: Is the Urdu Version of Mini-BESTest a Reliable and Valid Tool for Assessing the Dynamic Balance Impairments of Patients With Parkinson's Disease?
Brief Title: Reliability and Validity of Urdu Version of Mini-BESTest in Persons With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00275
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Balance
Keywords: Balance; Mini-BESTest; Parkinson's ; reliability; validity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Various clinical scales are available to investigate balance impairment, Mini-BESTest is one of them. Thus, this study aims to translate the Mini-BESTest into Urdu and investigate its psychometric properties in the Pakistani Parkinson's population with dynamic balance impairment.

DETAILED DESCRIPTION:
The aim of study is to translate and culturally adapt Mini-BESTest into Urdu language and secondly to investigate the reliability and validity of Urdu Version of Mini-BEStest in Parkinson's Pakistani population. This study will be cross sectional survey study in which convenience sampling technique will be used.

The results of study will help to know the validity and reliability of Mini-BESTest in Urdu version with dynamic balance impairments in Parkinson's population. The reliability of the scale will be checked through internal consistency and test-retest methods. Internal consistency will be analyzed with Cronbach's alpha value. Test-retest reliability will be assessed using an intraclass correlation coefficient with 80 patients.

ELIGIBILITY:
Inclusion Criteria:

1. All persons with Parkinson disease and ability to follow commands were included in the study.
2. living independently in the community
3. able to walk 6 m independently
4. willing to participate in the study.

Exclusion Criteria:

1. History of other neurological disorders
2. Musculoskeletal damage which affects walking ability
3. Presence of serious medical condition
4. History of surgical treatments for Parkinson disease
5. Not willing to participate in the study
6. history of faint, vertigo, dizziness,or taking medications which can cause dizziness
7. history of any medical condition which can affect balance.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The incidence of Parkinson disease increases by age especially after the age of 60 As we know equilibrium and postural control are essential for everyday work so postural instability, freezing of gait, impaired anticipatory and reactive balance, impaired cognition ,reduced leg muscle strength, reduced proprioception, and frontal lobe impairment are major cause of balance impairment and falls in persons with Parkinson disease and falling puts persons with Parkinson disease at a higher risk of fractures, soft tissue injury, immobilization, depression, daily activity restriction, and mortality
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Mini-BESTest Scale | 1st day
  A measuring instrument for the evaluation of dynamic balance is the Mini-BESTest Scale. Each item is scored from 0 to 2 , higher score 2 means better balance performance and 0 showing worst balance performance . Mini-BESTest 28 is the highest result possible
Berg Balance Scale | 1st day
  The Berg Balance Scale is an objective assessment of balance performance based on 14 items common to everyday activities. It is a 14 items scale that rates 0 (unable to perform) to 4 (normal performance) for each item. The total score is 56 points. Higher score higher balance ability.
Brief -BESTest Scale | 1st day
  The Brief -BESTest Scale is a shorter version of the BEStest Scale and takes less time to administer. It consist of eight items from six section . Each item is scored from 0 to 3, higher score means better balance performance. All items scores are summed to obtain the total score which ranges from 0 to 24.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No